CLINICAL TRIAL: NCT03694990
Title: Prospective Quality of Life Study in Pituitary Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jose Mattos, MD, Principal Investigator, University of Virginia
Other Study IDs: 20758
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Post Operative Care; Endoscopic Skull Base Surgery; Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Short-term: Patients will be scheduled for PO follow-up visits 2 weeks, and 8 weeks after surgery.
  Interventions: Other: Follow-up schedule
- Intermediate: Patients will be scheduled for PO follow-up visits 4 weeks, and 8 weeks after surgery.
  Interventions: Other: Follow-up schedule
- Long-term: Patients will be scheduled for PO follow-up visits 8 weeks after surgery.
  Interventions: Other: Follow-up schedule

INTERVENTIONS:
Other: Follow-up schedule — Patients will be randomized into 1 of 3 follow-up schedules for post-operative clinic visits.

SUMMARY:
Post-operative assessment and debridement are key components in patient care for surgery patients. However, a standardized protocol for management after endoscopic skull base surgery is unavailable. In this study, investigators will observe the effect of various follow-up schedules on the patient's quality of life after surgery. Patients who received surgery for pituitary adenoma will be placed randomly in 1 of 3 groups (short-term = follow-up in 2 weeks and 8 weeks after surgery; intermediate = 4 weeks and 8 weeks; long-term = 8 weeks). At each visit, patients will be asked to complete a packet of surveys and questionnaires that provide metrics on their quality of life in addition to receiving standard patient care (post-operative assessment and nasal debridement). Researchers hope to find that a follow-up schedule that has patients visiting the clinic closer to their surgery date will increase the patient's quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has surgery for pituitary adenoma at UVA after May 1st, 2018
* Has sellar and parasellar pathology
* ≥ 18 years old
* Can complete all parts of study in English

Exclusion Criteria:

* Extended approaches
* Use of naso-septal flap during the current surgical procedure
* Septoplasty
* Prior history of Chronic Rhinosinusitis (CRS)
* Prior history of sphenoidotomy
* < 18 years old
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving surgery for pituitary adenoma at UVA after May 1st, 2018.
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 survey scores for pre-op/initial visit | Survey results will be collected during the pre-op/initial 1 day visit
  Patient responses to the SNOT-22 will be collected and calculated.
SNOT-22 survey scores for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the SNOT-22 will be collected and calculated.
SNOT-22 survey scores for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the SNOT-22 will be collected and calculated.
SNOT-22 survey scores for 3-month contact | 3-month contact
  Patient responses to the SNOT-22 will be collected and calculated.
SNOT-22 survey scores for 6-month follow-up visit | 6-month post-op
  Patient responses to the SNOT-22 will be collected and calculated.
Anterior Skull Base QOL survey scores for pre-op/initial visit | collected during the pre-op/initial 1 day visit
  Patient responses to the Anterior Skull Base QOL will be collected and calculated.
Anterior Skull Base QOL survey scores for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the Anterior Skull Base QOL will be collected and calculated.
Anterior Skull Base QOL survey scores for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the Anterior Skull Base QOL will be collected and calculated.
Anterior Skull Base QOL survey scores for 3-month contact | 3-month contact
  Patient responses to the Anterior Skull Base QOL will be collected and calculated.
Anterior Skull Base QOL survey scores for 6-month follow-up visit | 6-month post-op
  Patient responses to the Anterior Skull Base QOL will be collected and calculated.
Pain Catastrophizing Scale (PCS) response for pre-op/initial visit | collected during the pre-op/initial 1 day visit
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Pain Catastrophizing Scale (PCS) response for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Pain Catastrophizing Scale (PCS) response for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Pain Catastrophizing Scale (PCS) response for 3-month contact | 3-month contact
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Pain Catastrophizing Scale (PCS) response for 6-month follow-up visit | 6-month post-op
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Questionnaire of Olfactory Disorders survey scores for pre-op/initial visit | collected during the pre-op/initial 1 day visit
  Patient responses to the Pain Catastrophizing Scale (PCS) will be collected and calculated.
Questionnaire of Olfactory Disorders survey scores for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the Questionnaire of Olfactory Disorders will be collected and calculated.
Questionnaire of Olfactory Disorders survey scores for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the Questionnaire of Olfactory Disorders will be collected and calculated.
Questionnaire of Olfactory Disorders survey scores for 3-month contact | 3-month contact
  Patient responses to the Questionnaire of Olfactory Disorders will be collected and calculated.
Questionnaire of Olfactory Disorders survey scores for 6-month follow-up visit | 6-month post-op
  Patient responses to the Questionnaire of Olfactory Disorders will be collected and calculated.
Skull Based Inventory scores for pre-op/initial visit | collected during the pre-op/initial 1 day visit
  Patient responses to the Skull Based Inventory will be collected and calculated.
Skull Based Inventory scores for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the Skull Based Inventory will be collected and calculated.
Skull Based Inventory scores for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the Skull Based Inventory will be collected and calculated.
Skull Based Inventory scores for 3-month contact | 3-month contact
  Patient responses to the Skull Based Inventory will be collected and calculated.
Skull Based Inventory scores for 6-month follow-up visit | 6-month post-op
  Patient responses to the Skull Based Inventory will be collected and calculated.
Quality of Recover (QOR 40) survey scores for pre-op/initial visit | collected during the pre-op/initial 1 day visit
  Patient responses to the Quality of Recover (QOR 40) will be collected and calculated.
Quality of Recover (QOR 40) survey scores for 2-week or 4-week follow-up visit | 2-weeks or 4-weeks after surgery (based on group)
  Patient responses to the Quality of Recover (QOR 40) will be collected and calculated.
Quality of Recover (QOR 40) survey scores for 8-week follow-up visit | 8-weeks post-op
  Patient responses to the Quality of Recover (QOR 40) will be collected and calculated.
Quality of Recover (QOR 40) survey scores for 3-month contact | 3-month contact
  Patient responses to the Quality of Recover (QOR 40) will be collected and calculated.
Quality of Recover (QOR 40) survey scores for 6-month follow-up visit | 6-month post-op
  Patient responses to the Quality of Recover (QOR 40) will be collected and calculated.

SECONDARY OUTCOMES:
Physician's notes/Patient progress notes for patient clinic visits | Clinic visit notes and/or patient progress notes will be collected during the pre-op/initial 1 day visit, subsequent follow-up visits (2-weeks, 4-weeks, and 8-weeks post-op), and final visit (6-months post-op).
  Notes taken by the physician/medical staff during subject's clinic visit (i.e. lesion pathology, cavernous sinus invasion, suprasellar extension, post-op assessment, presence of nasal synechiae, rate of medpor graft extrusion)
Endoscopy scores | Endoscopy scores will be collected during the pre-op/initial 1 day visit, subsequent follow-up visits (2-weeks, 4-weeks, and 8-weeks post-op), and final visit (6-months post-op).
  Lund-Kennedy scoring of endoscopic imaging of nasal cavity
Surgery notes/outcomes | intraoperative
  Surgeon's notes on subject surgery (i.e. occurrence of intra-operative leak, type of packing used)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Mattos, MD, Principal Investigator — University of Virginia School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tien DA, Stokken JK, Recinos PF, Woodard TD, Sindwani R. Comprehensive Postoperative Management After Endoscopic Skull Base Surgery. Otolaryngol Clin North Am. 2016 Feb;49(1):253-63. doi: 10.1016/j.otc.2015.09.015. PMID 26614842
- [Background] Nyquist GG, Rosen MR, Friedel ME, Beahm DD, Farrell CJ, Evans JJ. Comprehensive management of the paranasal sinuses in patients undergoing endoscopic endonasal skull base surgery. World Neurosurg. 2014 Dec;82(6 Suppl):S54-8. doi: 10.1016/j.wneu.2014.07.027. PMID 25496636
- [Background] Suberman TA, Zanation AM, Ewend MG, Senior BA, Ebert CS Jr. Sinonasal quality-of-life before and after endoscopic, endonasal, minimally invasive pituitary surgery. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):161-6. doi: 10.1002/alr.20029. Epub 2011 Apr 26. PMID 22287366
- [Background] Little AS, Kelly DF, Milligan J, Griffiths C, Prevedello DM, Carrau RL, Rosseau G, Barkhoudarian G, Jahnke H, Chaloner C, Jelinek KL, Chapple K, White WL. Comparison of sinonasal quality of life and health status in patients undergoing microscopic and endoscopic transsphenoidal surgery for pituitary lesions: a prospective cohort study. J Neurosurg. 2015 Sep;123(3):799-807. doi: 10.3171/2014.10.JNS14921. Epub 2015 Apr 17. PMID 25884256
- [Background] Woodmansee WW, Carmichael J, Kelly D, Katznelson L; AACE Neuroendocrine and Pituitary Scientific Committee. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY DISEASE STATE CLINICAL REVIEW: POSTOPERATIVE MANAGEMENT FOLLOWING PITUITARY SURGERY. Endocr Pract. 2015 Jul;21(7):832-8. doi: 10.4158/EP14541.DSCR. PMID 26172128